CLINICAL TRIAL: NCT04428788
Title: A Phase 1, Multi-center, Open-label, Dose Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Cc-94676 in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: Study to Evaluate the Safety and Tolerability of CC-94676 in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-94676-PCA-001; U1111-1251-9174 (Other: WHO)
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; CC-94676; Castration-resistant prostate cancer; Adenocarcinoma of the prostate; Prostatic Neoplasms Castration-Resistant; Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-94676, CC1083611, and CC1083610 (Experimental)
  Interventions: Drug: CC-94676; Drug: CC1083611; Drug: CC1083610

INTERVENTIONS:
Drug: CC-94676 — Specified dose on specified days
  Other Names: BMS-986365
Drug: CC1083611 — Specified dose on specified days
  Other Names: BMS-986409
Drug: CC1083610 — Specified dose on specified days
  Other Names: BMS-986410

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary efficacy of CC-94676 in men with progressive metastatic castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Progressed on androgen deprivation therapy (ADT) and at least one prior secondary hormonal therapy approved for castration-resistant prostate cancer (CRPC)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Prior treatment with an androgen receptor (AR) degrader
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 1 year prior to the first dose of IP
* Clinically significant venous thromboembolism within 3 months prior to the first dose of IP
* Any significant medical condition, such as uncontrolled infection, laboratory abnormality, or psychiatric illness

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) evaluated using the NCI CTCAE v5.0 criteria | From the time of consent at screening until 28 days after thesubject discontinues study treatment.
Dose-limiting toxicity (DLT) | Up to 35 days
Non-tolerated dose (NTD) | Up to 35 days
Maximum tolerated dose (MTD) | Up to 35 days

SECONDARY OUTCOMES:
Confirmed Prostate Specific Antigen (PSA) decline of ≥ 50% from baseline (PSA50) | Up to approximately 4 years
Objective soft tissue response defined by complete response (CR) or partial response (PR) per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) | Up to approximately 4 years
Duration of response (DOR) | Up to approximately 4 years
Proportion of participants alive and not progressed at 6 months | Up to 6 months after treatment is discontinued
PSA Progression Free Survival (PFS) | Up to approximately 4 years
Radiographic progression free survival (rPFS) | Up to approximately 4 years
Overall survival (OS) | Up to approximately 4 years
Overall Survival (OS) rate summarized using the Kaplan-Meier method for the treated population | Up to approximately 4 years
Pharmacokinetics - Area under the plasma concentration time curve (AUC) | Up to 35 days
Pharmacokinetics - Maximum plasma concentration (Cmax) | Up to 35 days
Pharmacokinetics - Time to Cmax (Tmax) | Up to 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (19):
  - Local Institution - 116, Stanford, California
  - Local Institution - 122, Washington D.C., District of Columbia
  - Local Institution - 103, Sarasota, Florida
  - Local Institution - 121, Thomasville, Georgia
  - Local Institution - 108, Baltimore, Maryland
  - Local Institution - 104, Boston, Massachusetts
  - Local Institution - 117, Ann Arbor, Michigan
  - Local Institution - 102, Grand Rapids, Michigan
  - Local Institution - 112, New York, New York
  - Local Institution - 109, New York, New York
  - Local Institution - 105, New York, New York
  - Local Institution - 106, Durham, North Carolina
  - Local Institution - 120, Allentown, Pennsylvania
  - Local Institution - 113, Philadelphia, Pennsylvania
  - Local Institution - 107, Dallas, Texas
  - Local Institution - 119, Houston, Texas
  - Local Institution - 101, San Antonio, Texas
  - Local Institution - 115, Seattle, Washington
  - Local Institution - 111, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com